CLINICAL TRIAL: NCT02145715
Title: A Phase I/IIa Trial of VTD-panobinostat Treatment and Panobinostat Maintenance in Relapsed and Relapsed/Refractory Multiple Myeloma Patients
Brief Title: Velcade, Thalidomide, Dexamethasone and Panobinostat Treatment and Panobinostat Maintenance in Multiple Myeloma
Acronym: MUKsix
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Prof Jamie Cavenagh (Other)
Collaborators: Myeloma UK (Other); Novartis (Industry)
Responsible Party: Sponsor-Investigator, Prof Jamie Cavenagh, Chief Investigator, University of Leeds
Organization: University of Leeds (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM12/10174
Record Dates: First submitted 2013-03-01; First posted 2014-05-23 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Thalidomide; Dexamethasone; Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Velcade, Thalidomide, Dexamethasone (VTD) + Panobinostat (Experimental): Up to 16 cycles of VTD+Panobinostat followed by panobinostat maintenance for 1 year or until disease progression.
  * Induction - Cycles 1-16 (21-day cycle)
    * Velcade: 1.3mg/m2 (subcutaneous) on days 1 and 8
    * Thalidomide: 100mg (PO)on days 1 -21
    * Dexamethasone: 20 mg (PO) on days 1, 2, 8 and 9
    * Panobinostat: 10mg, 15mg or 20mg days 1, 3, 5, 8, 10 and 12 Dose depends on cohort entry at registration during the dose escalation phase. The recommended dose will be used during the expansion phase.
  * Panobinostat monotherapy maintenance for 1 year. Panobinostat will be given at the same dose as the recommended dose during expansion phase
  Interventions: Drug: Velcade; Drug: Thalidomide; Drug: Dexamethasone; Drug: Panobinostat

INTERVENTIONS:
Drug: Velcade
  Other Names: Bortezomib
Drug: Thalidomide
Drug: Dexamethasone
Drug: Panobinostat

SUMMARY:
Velcade (bortezomib), thalidomide and dexamethasone (VTD) has been demonstrated to be a highly effective combination in both patients with previously untreated and those with relapsed multiple myeloma. In previously untreated patients VTD demonstrated clear superiority to TD as induction therapy prior to planned tandem autologous stem cell transplant.

The rationale of this trial is to combine a 'gold standard' antiMM combination with the HDAC inhibitor Panobinostat. There is emerging data to support the concept of clinical synergy between BTZ and HDACi's.

The purpose of this study is to determine the maximum tolerated dose (MTD) and estimated response rates of panobinostat, administered in combination with VTD, in subjects with relapsed and relapsed/refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a previous diagnosis of multiple myeloma based on IMWG 2003 definitions:

  * Monoclonal immunoglobulin (M component) on electrophoresis, and on immunofixation of serum or of total 24 hour urine
  * Bone marrow (clonal) plasma cells ≥ 10% or biopsy proven plasmacytoma
  * Related organ or tissue impairment (CRAB symptoms, anemia, hypercalcemia, lytic bone lesions, renal insufficiency, hyperviscosity, amyloidosis or recurrent infections)
* Relapsed and relapsed-and-refractory myeloma who have received 1-4 prior lines and now require further treatment
* Able to give informed consent and willing to follow study protocol
* Aged 18 years or over
* ECOG Performance Status ≤2
* Required laboratory values within 14 days of registration:

  * Absolute neutrophil count ≥1.0 x 109/L.
  * Platelet count ≥100 x 109/L.
  * Haemoglobin ≥8.0g/dL.
  * Bilirubin ≤2 upper limit of normal (ULN)
  * AST and/or ALT ≤2.5 ULN; except in subjects with known hepatic involvement, where AST and/or ALT ≤5.0 ULN
  * Serum creatinine ≤2.0 ULN
  * Corrected calcium ≤2.8 mmol/L.
* Anticipated survival of at least 3 months
* Evaluable disease per modified IWG criteria, utilising the following assessments as appropriate:

  * Serum M protein ≥ 10g/l.
  * Urine M protein ≥ 200mg/24 hours
  * Serum free light chain assay: involved FLC level ≥ 100mg/l. Provided serum FLC ratio is abnormal
* Female subjects of child-bearing potential must have a negative pregnancy test at baseline and agree to use dual methods of contraception for the duration of the study and must continue to do so for 3 months after the end of treatment. Male subjects must agree to use a barrier method of contraception for the duration of the study if sexually active with a female of child-bearing potential and must continue to do so for 3 months after the end of treatment.

Exclusion Criteria:

* Pregnant (positive pregnancy test) or breastfeeding women.
* Non-secretory Multiple Myeloma Previous anti-tumour therapies, including prior experimental agents or approved anti-tumour small molecules and biologics, within 28 days before the start of protocol treatment. Steroid therapy is permitted (maximum 160 mg dexamethasone or equivalent), but must be stopped 48 hours prior to study drug administration. Bisphosphonates for bone disease and radiotherapy for palliative intent are also permitted.
* Concurrent or previous malignancies (<12 months post end of treatment) at other sites with the exception of appropriately treated localised epithelial skin or cervical cancer, or incidental histologic findings of prostate cancer (TMN stage T1a or 1b). Patients with histories (≥12 months) of other tumours may be entered.
* Poorly controlled or serious medical or psychiatric illness that, in the Investigator's opinion, is likely to interfere with participation and/or compliance in this clinical study
* Patients with significant cardiovascular disease (e.g. history of congestive heart failure requiring therapy, presence of severe valvular heart disease, presence of an atrial or ventricular arrhythmia requiring treatment, uncontrolled hypertension, a history of clinically significant QTc abnormalities)
* Active symptomatic fungal, bacterial, and/or viral infection including known active HIV or known viral (A, B, or C) hepatitis.
* Gastrointestinal disorders that may interfere with absorption of the study drug
* Patients who have been refractory to prior bortezomib, i.e. did not achieve at least an MR, or who have progressed on therapy or within 60 days of last dose
* Participants with peripheral neuropathy CTC grade 2 or higher or grade 1 with pain within 14 days prior to registration
* Any history or known hypersensitivity to any of the study medications or excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-07 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) | From cycle 1 day 1 up to the administration of cycle 2 day 1 (up to 22 days)
  The number of participants experiencing DLTs within the first cycle of VTD-pano will be presented, with descriptive summaries of the specific DLTs observed. Summaries will be presented for each dose level.
Proportion o f participants achieving at least partial response | within 16 cycles of therapy (an expected average of 48 weeks)
  The proportion of participants achieving at least a partial response within 16 cycles of VTD-pano will be presented, with corresponding 80% and 95% confidence intervals

SECONDARY OUTCOMES:
Safety and toxicity | Throughout the trial, expected to be 3 years
  The proportion of participants experiencing DLTs and other toxicities, overall and by cycle as graded by CTCAE V4.0.
Proportion of patients with each maximum response category | within 16 cycles of therapy (an expected average of 48 weeks)
  The number and proportion of participants in each response category within 16 cycles of VTD-pano will be presented with corresponding 95% confidence intervals.
Time to maximum response to therapy | from registration until the participant achieves any of the categories CR, VGPR, PR, MR or SD as their maximum response (up to 100 weeks - 48 weeks of treatment plus 52 weeks maintenance)
  Time to maximum response is defined as the time from registration until the patient achieves any of the categories CR, VGPR, PR, MR or SD as their maximum response. Median time to maximum response will be presented.
Progression free survival | from registration to first documented evidence of disease progression or death (up to 100 weeks)
  A progression-free survival curve will be calculated using the Kaplan Meier method and median PFS estimates will be presented.
Compliance to therapy | from initial treatment received as per protocol until treatment withdrawal (up to 100 weeks)
  Compliance to therapy will be summarised descriptively, including number of doses missed and number of dose reductions throughout the treatment period.
Feasibility of panobinostat maintenance | up to 12 months
  The duration of maintenance and reasons for stopping will be summarised
Overall survival | from registration to date of death
  Overall survival (OS) curves will be calculated using the Kaplan Meier method. Median OS, and OS estimates at 12 months, will be presented, if appropriate.
The proportion of participants mobilising sufficient stem cells for transplant(out of those undergoing mobilisation) | up to 16 cycles of therapy (an expected average of 48 weeks)
  To be determined by the satisfactory collection of sufficient numbers of stem cells to support high-dose chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Cavenagh, MRCPath, Principal Investigator — St. Bartholomew's Hospital
Locations (5):
- United Kingdom (5):
  - Birmingham Heartlands Hospital, Birmingham, UK
  - Royal Liverpool University Hospital, Liverpool
  - St Bartholomew's Hospital, London
  - University College London Hospitals NHS Foundation Trust, London
  - Guy's Hospital, London

REFERENCES:
- [Derived] Popat R, Brown SR, Flanagan L, Hall A, Gregory W, Kishore B, Streetly M, Oakervee H, Yong K, Cook G, Low E, Cavenagh J; Myeloma UK Early Phase Clinical Trial Network. Bortezomib, thalidomide, dexamethasone, and panobinostat for patients with relapsed multiple myeloma (MUK-six): a multicentre, open-label, phase 1/2 trial. Lancet Haematol. 2016 Dec;3(12):e572-e580. doi: 10.1016/S2352-3026(16)30165-X. Epub 2016 Nov 12. PMID 27843120